CLINICAL TRIAL: NCT03385226
Title: Phase II Trial of Pembrolizumab and Radiotherapy in Cutaneous T-cell Lymphoma
Brief Title: A Trial Assessing the Effect of Pembrolizumab Combined with Radiotherapy in Patients with Relapsed, Refractory, Specified Stages of Cutaneous T-cell Lymphoma (CTCL) Mycosis Fungoides (MF)/Sezary Syndrome (SS)
Acronym: PORT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/17/0053; 2017-000433-30 (EudraCT Number)
Record Dates: First submitted 2017-12-12; First posted 2017-12-28 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Cutaneous T Cell Lymphoma; Mycosis Fungoides/Sezary Syndrome
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Recurrence | interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab with radiotherapy (Experimental): All patients will receive
  * single 200mg pembrolizumab IV infusions given 3-weekly until 2 years post study entry, termination of treatment, disease progression or unacceptable toxicity
  * radiotherapy, 12Gy in 3 fractions
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a humanised monoclonal antibody which targets the programmed cell death 1 (PD-1) receptor. It blocks a protective mechanism on cancer cells, and allows the immune system to destroy those cancer cells.
  Other Names: Chemical Abstract Service (CAS) number - 1374853-91-4
Radiation: Radiotherapy — 12Gy in 3 fractions

SUMMARY:
Trial Subjects (patients), will receive single infusions of pembrolizumab every 3 weeks until disease progression or unacceptable toxicity develops. They will receive radiotherapy at week 12.

DETAILED DESCRIPTION:
Trial Subjects (patients) who are deemed eligible for the trial will be administered a single infusion of pembrolizumab (200mg) every 3 weeks. At week 12, patients will be planned to start radiotherapy at a dose of 12 Gray (Gy) in 3 fractions which will be given concomitantly with pembrolizumab. Patients who progress on pembrolizumab before week 12 will start radiotherapy as soon as possible after progression. Following completion of radiotherapy, patients will continue receiving pembrolizumab at 3 weekly intervals for a maximum of 2 years until disease progression or unacceptable toxicity develops. Patients on pembrolizumab will be seen every 3 weeks until 2 years after study entry, while Patients who progressed/ stopped pembrolizumab will be seen annually for survival/disease status only. Patients completing 2 years of treatment will then be followed up annually for survival and disease status until the end of trial is declared (2 years after the last patient is registered).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of Stage IB-IVB CTCL mycosis fungoides (MF)/Sézary Syndrome (SS)
* Have relapsed, are refractory or progressed after at least 1 systemic therapy
* Skin biopsy at the time of or within 6 months prior to study entry
* Patients must have a total mSWAT (modified Severity Weighted Assessment Tool) score of ≥10 OR have 2 or more measurable tumours of any size. Of this area: there should be at least 1 cutaneous lesion (MF) or a defined area of involved skin (erythrodermic MF or SS) which is an appropriate target for palliative radiotherapy. There should be an area of skin involved by measurable Mycosis Fungoides/SS that will not be irradiated (To assess the abscopal effect of radiotherapy)
* Have a minimum wash-out and adverse event (AE) recovery period from previous treatments (e.g. topical therapy, phototherapy, local radiotherapy, monoclonal antibody, systemic cytotoxic anticancer treatment or other novel agents) prior to the first dose of pembrolizumab
* Have ECOG performance status of 0 or 1
* Life expectancy of at least 6 months
* Demonstrate adequate organ function
* Female patients of childbearing potential must have a negative urine or serum pregnancy test at pre-registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Willing to comply with the contraception requirements
* Written informed consent

  •Exclusion Criteria:
* Received chemotherapy or targeted small molecule therapy within 4 weeks prior to study entry or has not recovered from adverse events due to agents administered >4 weeks earlier (except patients with ≤ grade 2 neuropathy)
* Is currently or has participated in an IMP or device study within 4 weeks prior to the first dose of pembrolizumab
* Received any other monoclonal antibody within 15 weeks prior to the first dose of pembrolizumab or has not recovered (≤ grade 1 or to baseline level) from adverse events due to agents administered >4 weeks earlier. The exception to this is alemtuzumab which should not have been administered in the previous 12 weeks
* Additional malignancy that is progressing or requires active treatment
* Patients with known central nervous system (CNS) involvement with lymphoma
* Hypersensitivity to pembrolizumab or its excipients
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Stable use of corticosteroids (at a dose no higher than 10mg prednisolone per day over the preceding 4 weeks) is allowed
* Diagnosis of prior immunodeficiency or organ-transplant requiring immunosuppressive therapy
* Current or prior use of immunosuppressive therapy within 7 days prior to start of treatment except the following: intranasal, inhaled, topical steroids or local steroid injections (eg. Intra-articular injection); systemic corticosteroids at physiologic doses (10mg/day or less of prednisolone or equivalent)
* Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2 therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia
* Has known history of, or any evidence of active, non-infectious pneumonitis
* History of other pulmonary disease such as interstitial lung disease, emphysema or chronic obstructive pulmonary disease
* Is pregnant or breastfeeding
* Has a known history of active TB
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial or interfere with the subject's participation for the full duration of the trial or to participate in the trial is not in the patient's best interest, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with the requirements of the trial
* Has a known history of HIV
* Has known active Hepatitis B or Hepatitis C
* Has received a live vaccine within 30 days prior to the planned start of study medication
* Patients who have previously received a solid organ transplant
* Patients who have previously received any allogeneic transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response (Global Assessment) | 24 weeks after commencement of pembrolizumab
  Overall Response of the combination of pembrolizumab plus radiotherapy

SECONDARY OUTCOMES:
Response | 12 weeks after start of pembrolizumab
  Response at the 5th infusion of pembrolizumab, typically 12 weeks after start of treatment
Change in Global Response | 24 weeks after start of pembrolizumab
  Change in Global Response from the 5th infusion to the 9th infusion, typically from week 12 to week 24
Safety and toxicity | 5 months after last dose of pembrolizumab (anticipated 2 years and 5 months after last patient being registered)
  Number & Percentage of patients who suffer grade 3 or 4 toxicity
Response Duration | Time from date of first confirmed response to the first date of diagnosis of progressive disease or death from any cause (anticipated by 2 years and 5 months after the last patient being registered)
  Duration of tumour response
Progression Free Survival | Time from date of registration to the date of first progression or death from any cause ((anticipated by 2 years and 5 months after the last patient being registered)
  Disease progression or death
Overall Survival | Time from date of registration to the date of death from any cause ((anticipated by 2 years and 5 months after the last patient being registered)
  Death
Number of patients achieving abscopal effect | Through study completion, 2 years post last patient being registered

OTHER OUTCOMES:
Assessment of changes in the immune status | 24 weeks after start of pembrolizumab
  Peripheral blood mononuclear cell phenotyping
Analysis of plasma High Mobility Group Box 1 (HMGB-1) isoform levels | 24 weeks after start of pembrolizumab
  Peripheral blood mononuclear cell phenotyping
Functional analysis of isolated cell populations | 24 weeks after start of pembrolizumab
  Peripheral blood mononuclear cell phenotyping
Assessment of diversity and clonality of T cell clones | 24 weeks after start of pembrolizumab
  DNA extraction for T cell receptor sequencing
Evaluation of immune signatures for responders and non-responders | 24 weeks after start of pembrolizumab
  Peripheral blood mononuclear cell phenotyping
Epitope screening for tumour infiltrating lymphocyte specific neo-antigens | 24 weeks after start of pembrolizumab
  Peripheral blood mononuclear cell phenotyping
Immunohistochemical analysis of expression of immunological checkpoints | At baseline
  Assessment of PD-L1 expression
Investigation of the baseline tumour immune microenvironment | At baseline
  Immune cell infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Tim Illidge, Principal Investigator — University of Manchester
Locations (11):
- United Kingdom (11):
  - University Hospital Birmingham, Birmingham
  - Velindre Cancer Centre, Cardiff
  - University Hospital Coventry, Coventry
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guy's & St Thomas', London
  - The Christie, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Freeman Hospital, Newcastle
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Southampton University Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Narducci MG, Tosi A, Frezzolini A, Scala E, Passarelli F, Bonmassar L, Monopoli A, Accetturi MP, Cantonetti M, Antonini Cappellini GC, De Galitiis F, Rosato A, Picozza M, Russo G, D'Atri S. Reduction of T Lymphoma Cells and Immunological Invigoration in a Patient Concurrently Affected by Melanoma and Sezary Syndrome Treated With Nivolumab. Front Immunol. 2020 Sep 25;11:579894. doi: 10.3389/fimmu.2020.579894. eCollection 2020. PMID 33072126